CLINICAL TRIAL: NCT06737224
Title: The Impact of a 48-hour Fast with or Without Exercise on Immune Cell Function, Bioenergetics, and Glycemic Control in Healthy Active Adults: a Randomized Crossover Trial
Brief Title: The Impact of a 48-hour Fast with or Without Exercise on Immune Cell Metabolism and Glycemic Control in Healthy Active Adults
Acronym: FASTEX
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Jonathan Little, Professor, University of British Columbia
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: H24-01732
Record Dates: First submitted 2024-10-08; First posted 2024-12-17 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-03

CONDITIONS: Fasting; Immune Function; Glucose Tolerance
Keywords: Exercise; Immunometabolism; Glycemic control
MeSH Terms: conditions — Fasting; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized crossover, within-subject, repeated measures
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fasting + Exercise (FAST+EX): fasting + exercise condition (Experimental): 48-hour fast with 60 minutes of cycling on the first and second day of the fast.
  Interventions: Other: Fasting + Exercise (FAST+EX): fasting + exercise condition
- Fasting only (FAST): Non-exercise fasting condition (Experimental): 48-hour fast with no structured exercise on fasting days.
  Interventions: Other: Fasting only (FAST): Non-exercise fasting condition

INTERVENTIONS:
Other: Fasting + Exercise (FAST+EX): fasting + exercise condition — Participants will complete a 48-hour fast. One hour of exercise will be performed on each morning of the fast.
  Arms: Fasting + Exercise (FAST+EX): fasting + exercise condition
Other: Fasting only (FAST): Non-exercise fasting condition — Participant will complete a 48-hour fast. No structured exercise will be performed during each of the fasting days.
  Arms: Fasting only (FAST): Non-exercise fasting condition

SUMMARY:
Many individuals engage in fasting for its purported health benefits but the effects of fasting on immune cell and whole body metabolism are not well understood in humans. Moreover, how exercising during a prolonged fast impacts immunometabolic outcomes is unclear. This study will determine how a 2 day fast - performed with or without daily exercise - impacts immune cell bioenergetics, immune cell function, and whole-body glycemic control in healthy active individuals.

DETAILED DESCRIPTION:
Participants will perform two, 48-hour fasts separated by 5 days while wearing a continuous glucose monitor to measure glycemic responses. The order of the trials will be randomized for each participant. The two trials will include an exercise condition (FAST+EX) and a control, non-exercise condition (FAST). During the FAST+EX trial, participants will perform 60 minutes of cycling on each of the two days of the fast. Each bout of exercise will be 60 minutes in duration and consist of 50 minutes of cycling at 60% of predicted heart rate reserve (HRR) followed by 5 x 1-minute intervals at 90% of predicted HRR with 1-minute of passive recovery between each interval. During the FAST trial, participants will be asked to refrain from any structured exercise during the days of the fast. To start the trial, participants will arrive at the lab following an overnight fast. They will consume a standardized meal replacement (Ensure Plus Calories) and blood will be drawn 2 hours post-ingestion. Participants will come to the lab 24 and 48 hours later for subsequent blood draws prior to breaking their fast with the same standardized meal replacement. Another blood sample will be taken 2 hours post-prandial. Participants will be asked to replicate food consumption in each condition for the 24-hour period after they break their fast, and consume the same standardized meal replacement on the morning following the completion of each fast to measure free-living glycemic control 24-hours after a fast performed with or without exercise. There will be a five-day wash out period in between the completion of both trials for all participants.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 19 and 35 years.
* Physically active (engaging in ≥150 minutes of weekly moderate to vigorous physical activity).

Exclusion Criteria:

* History of cardiometabolic diseases or inflammatory diseases (e.g., chronic obstructive pulmonary disease (COPD), rheumatoid arthritis, cardiovascular disease).
* Individuals currently following a ketogenic diet, low-calorie diet, periodic fasting regimen, or consuming ketogenic supplements (e.g., exogenous ketone drinks).
* Cigarette/vaping smoking.
* Physical limitation that will impair the ability of the participant to perform exercise.
* Individuals having a body mass index (BMI) over 30 kg/m2.
* Cancer diagnosis in the past 5 years.
* Taking anti-inflammatory drugs (e.g., ibuprofen, aspirin, naproxen).
* Being unable to read or communicate in English.

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Monocyte mitochondrial respiration | Baseline and 48 hours
  Mitochondrial respiration will be measured in primary human monocytes using high resolution respirometry before and after a 48-hour fast performed with or without exercise.

SECONDARY OUTCOMES:
Alteration in immune cell functions | Baseline and 48 hours
  Immune cell functions will be assessed with the combination of whole blood cultures treated with lipopolysaccharide (with or without interleukin-10) and the subsequent measurement of cytokine secretion, immune cell counts, and phenotyping via flow cytometry, both before and after 48 hours fast (with and without exercise).
Change in glucose tolerance | Baseline, after 48 hours of fasting, and 24 hours after breaking the fast in free-living condition)
  Investigate whether exercise performed during a 48-hour fast can reduce the temporary glucose intolerance typically seen after fasting, both in controlled and free-living conditions. Glucose tolerance will be evaluated by measuring capillary glucose levels before, and at 30, 60, and 120 minutes after a mixed meal tolerance test.
Blood pressure | Baseline, 24 hours into the fast, and at the end of the fast (48 hours)
  Systolic and diastolic blood pressure, as well as heart rate, will be measured using an automatic blood pressure device at baseline (Day 1), 24 hours into the fast (Day 2), and at the end of the 48-hour fast (Day 3) in both conditions (fasting alone and fasting with exercise).
Rate and level of ketosis | Baseline, 24 hours and 48 hours during fasting
  Examine whether performing exercise at the beginning and during a fast can influence the ketone levels achieved after 24 and 48 hours of fasting. Capillary beta-hydroxybutyrate (a ketone body) will be measured via finger pricks using the Freestyle Neo ketone test.
Compensatory movement behaviour | During and 48 hours after the fast
  Explore whether adding exercise during fasting could intensify compensatory movement behaviors, as indicated by changes in sedentary behavior, light physical activity, and moderate to vigorous physical activity, measured using an accelerometer (ActivPAL).
Hunger sensation | At baseline, 12:00, 18:00 during the first and second day of the fast.
  Hunger will be assessed using a 10-cm visual analogue scale at several time points: in the morning at the start of the fast, at 12:00 and 18:00 on the same day, at the same times the following day, and just before breaking the fast 48 hours later.
Sleep quality | Baseline the morning before starting the fast, after 24 hours of fasting, and again after 48 hours of fasting.
  Sleep quality will be assessed using a 10-cm visual analog scale based on the Richards-Campbell Sleep Questionnaire (2000). Measurements will be taken at baseline the morning before starting the fast, after 24 hours of fasting, and again after 48 hours of fasting.
Affect during exercise | Before, during (e.g., at 10, 20, 30, 40, and 50 minutes as well as during intervals 1,2,3,4, and 5 at the end of the intervals as well as during the passive recovery) and following the two exercises conditions (post 5 minutes in a seated position).
  The Feeling Scale (FS) developed by Hardy and Rejeski (Hardy & Rejeski, 1989) will be used to measure affective valence when exercise is performed in the fed (Baseline) and fasted state (24h fasted). Specifically, FS will be measured before, during (e.g., at 10, 20, 30, 40, and 50 minutes as well as during intervals 1,2,3,4, and 5 at the end of the intervals as well as during the passive recovery) and following the two exercises conditions (post 5 minutes in a seated position).
Remembered Enjoyment | 10 minutes after each exercise session.
  Remembered enjoyment will be measured with the original Physical Activity Enjoyment Scale (PACES; Kendzierski & DeCarlo, 1991) 10 minutes following each supervised exercise session (i.e., fed and fasted).
Rate of perceived exertion | During both exercise sessions at 10, 20, 30, 40, and 50 minutes as well as during intervals 1, 2, 3, 4, and 5 at the end of the intervals.
  Rate of perceived exertion will be measured during both exercise sessions (i.e., fed and fasted) at 10, 20, 30, 40, and 50 minutes as well as during intervals 1,2,3,4, and 5 at the end of the intervals.
Glucose homeostasis | During and 24 hours after both condition
  Glucose homeostasis will be evaluated using a continuous glucose monitor (Freestyle Libre 2, Abbott) under both conditions-fasting alone and fasting combined with exercise. Key markers of glucose homeostasis will be assessed based on Battelino et al. (2022; Lancet Diabetes Endocrinol), and will include average glucose levels, glycemic variability (SD), and time spent below (≤ 3.9 mmol/L), within (3.9-10.0 mmol/L), and above range (≥ 10.0 mmol/L).

CONTACTS AND LOCATIONS:
Locations (1):
- University of British Columbia Okanagan Campus, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared to ensure the privacy and confidentiality of participants, in accordance with ethical guidelines and data protection regulations. Additionally, this was not included in the informed consent, which did not cover data sharing or address potential risks of re-identification.